CLINICAL TRIAL: NCT02875795
Title: A Speech Disorders Severity Index to Measure the Impact of Oral and Pharyngeal Cavity on Speech Production
Brief Title: Carcinologic Speech Severity Index
Acronym: C2SI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: University Jean-Jaures, Toulouse, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14 7414 07
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Head and Neck Cancer
Keywords: linguistic; quality of life
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- speech intelligibility (Experimental): speech intelligibility is registered by an automatic speech processing tool
  Interventions: Procedure: automatic speech processing tool

INTERVENTIONS:
Procedure: automatic speech processing tool

SUMMARY:
The hypothesis of the present study is that an automatic assessment technic can measure the impact of the speech disorders on the communication abilities giving a severity index of speech in patients treated for head and neck and particularly for oral and pharyngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Oral and Pharyngeal cancer T2 to T4 for having a wide dynamic of deficit
* Treatment by surgery and/or radiotherapy and/or chemotherapy
* Delay after the end of the treatment of minimum 6 months.

Exclusion Criteria:

* Patients with a previous speech disorders (ie stuttering… )
* Patients not able to perform the whole task

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
carcinologic speech severity index | day 0
  The main objective is to demonstrate that the carcinologic speech severity index (C2SI), obtained by an automatic speech processing tool, produces equivalent or superior outcomes than a score of speech intelligibility obtained by human listeners, in terms of quality of life foreseeing the speech handicap, after the treatment of oral and/or pharyngeal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie WOISARD, Md, Principal Investigator — woisard.v@chu-toulouse.fr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Balaguer M, Boisguerin A, Galtier A, Gaillard N, Puech M, Woisard V. Assessment of impairment of intelligibility and of speech signal after oral cavity and oropharynx cancer. Eur Ann Otorhinolaryngol Head Neck Dis. 2019 Oct;136(5):355-359. doi: 10.1016/j.anorl.2019.05.012. Epub 2019 Jun 6. PMID 31178430